CLINICAL TRIAL: NCT05491642
Title: Study in Male / Postmenopausal Female Participants With Mild to Moderate Arterial Hypertension to Investigate Safety, Tolerability and Pharmacokinetics of Single and Multiple Doses of BAY 3283142 in a Randomized, Multi-center, Placebo-controlled, Single-blind, Group Comparison Design
Brief Title: A Study in Male and Female Participants (After Menopause) With Mild to Moderate High Blood Pressure to Learn How Safe the Study Treatment BAY3283142 is, How it Affects the Body and How it Moves Into, Through and Out of the Body After Taking Single and Multiple Doses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21592; 2022-001268-84 (EudraCT Number)
Record Dates: First submitted 2022-08-05; First posted 2022-08-08 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Chronic Kidney Disease; Hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Up-titration Scheme 1 (Experimental): Participants will receive 12 days treatment in total.
  Interventions: Drug: BAY3283142; Drug: Placebo to BAY3283142
- Up-titration Scheme 2 (Experimental): Participants will receive 12 days treatment in total.
  Interventions: Drug: BAY3283142; Drug: Placebo to BAY3283142
- Up-titration Scheme 3 (Experimental): Participants will receive 12 days treatment in total.
  Interventions: Drug: BAY3283142; Drug: Placebo to BAY3283142

INTERVENTIONS:
Drug: BAY3283142 — Oral administration
Drug: Placebo to BAY3283142 — Oral administration

SUMMARY:
Researchers are looking for a better way to treat people who have chronic kidney disease (CKD), a progressive decrease in the kidneys' ability to work properly.

In people with CKD, the kidneys do not remove wastes and extra fluid from the blood as well as they should. High blood pressure makes it more likely that the CKD gets worse.

The study treatment BAY3283142 is under development for treating CKD. It activates a protein called soluble guanylate cyclase (sGC) that generates cGMP - a molecule that relaxes blood vessels and is thought to have beneficial effects in CKD.

The participants do not benefit from this study. However, the study will provide information on how to use BAY3283142 in subsequent studies in people with CKD. As many people with CKD do also suffer from high blood pressure, this study is done in people with mild to moderate high blood pressure to safeguard the use of BAY3283142 in people with CKD in later studies.

The main purpose of this study is to learn how safe different single and multiple doses of the study treatment BAY3283142 are compared to placebo in male and female participants (after menopause) with mild to moderate high blood pressure. A placebo is a treatment that looks like a medicine but does not have any medicine in it.

To answer this, the researchers will compare the number of participants who have medical problems after taking BAY3283142 to those treated with placebo. Doctors keep track of all medical problems that happen in studies, even if they do not think they might be related to the study treatments.

Dependent on the treatment group, the participants will either take BAY3283142 or placebo as tablet once or twice a day. Patients will take one dose for 6 days and will then be switched to a higher dose for additional 6 days. In summary, three different dose combinations consisting of two different doses each will be tested.

Participants will be in the study for up to 7 weeks, including 12 treatment days (6 per dose step). They will stay in-house for 17 days starting two days before intake of the study treatment. In addition, one visit before and one visit after the in-house phase to the study site is planned.

During the study, the study team will:

* Check vital signs
* Take blood and urine samples
* Examine the participants' heart health using electrocardiogram (ECG)

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 30 to 78 years of age inclusive, at the time of signing the informed consent.
* Participants with diagnosis of mild to moderate systemic arterial hypertension receiving stable treatment for ≥8 weeks before the screening visit with not more than 2 antihypertensive drugs (note: 2 antihypertensive drugs combined within one pill count as 2 antihypertensive drugs).
* Mean systolic blood pressure (SBP) 120 - 160 mm Hg and mean diastolic blood pressure (DBP) 70-95 mm Hg at screening (mean out of triplicate measurements after supine rest for 15 min at screening).
* Estimated glomerular filtration rate (eGFR) ≥50 mL/min/1.73 m^2 (Chronic Kidney Disease Epidemiology Collaboration [CKD-Epi] formula) at screening and Study Day -2.
* Men and confirmed postmenopausal women.

Exclusion Criteria:

* Acute coronary syndrome (STEMI, NSTEMI, unstable angina, CABG, PCI, cardiac surgery).
* Ventricular tachycardia, atrial fibrillation, sick sinus syndrome, WPW syndrome.
* Thrombo-embolic events, e.g. stroke, TIA, deep vein thrombosis, pulmonary embolism.
* Systemic diseases: cancer (with the exception of appropriately treated basal cell carcinomas of the skin or uterine carcinoma in situ), autoimmune diseases (including also topically treated autoimmune diseases such as atopic dermatitis).
* Latent bleeding risk (diabetic retinopathy, history of gastrointestinal bleeding due to e.g. ulcers), inherited or acquired coagulopathies.
* Orthostatic intolerance in the modified standing blood pressure procedure at screening.
* Long-acting or short-acting nitrates or NO donors for any route including isosorbide dinitrate, isosorbide-5-mononitrate, pentaerythritol tetranitrate, nicorandil, nitrotriglyceride, molsidomin.
* Phosphodiesterase-5 (PDE-5) inhibitors or other soluble guanylate cyclase (sGC) stimulators or activators.
* Inhibitors of Uridine-5'-diphospho glucuronosyltransferase (UGT) 1A1, 1A3, 1A8 (e.g., probenecid) from 7 days before first study intervention until follow-up.
* Signs of hepatic dysfunction at the screening visit or at randomization as indicated by at least one of the following:

  * increases in isolated hepatic enzymes >1.3 fold ULN (alanine aminotransferase [ALT], aspartate aminotransferase [AST], alkaline phosphatase [AP], γ-GT).
  * Bilirubin > 1.3 fold ULN.

Ages: 30 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events per treatment arm | Up to 7 days after end of treatment with study intervention

SECONDARY OUTCOMES:
Area under the concentration versus time curve in a dosing interval (AUCτ) after single dose of BAY3283142 on Day 1 | Up to 24 hours post-dose
AUCτ after single dose of BAY3283142 on Day 1 divided by dose (AUCτ/D) | Up to 24 hours post-dose
Maximum observed drug concentration in measured matrix (Cmax) after single dose of BAY3283142 on Day 1 | Up to 24 hours post-dose
Cmax after single dose of BAY3283142 on Day 1 divided by dose (Cmax/D) | Up to 24 hours post-dose
AUC in a dosing interval after multiple doses of BAY3283142 on Day 12 (AUCτ,md) | Up to 24 hours post-dose
AUCτ,md after multiple doses of BAY3283142 on Day 12 divided by dose (AUCτ,md/D) | Up to 24 hours post-dose
Maximum observed drug concentration in measured matrix after multiple doses of BAY3283142 on Day 12 (Cmax,md) | Up to 24 hours post-dose
Cmax,md after multiple doses of BAY3283142 on Day 12 divided by dose (Cmax,md/D) | Up to 24 hours post-dose

CONTACTS AND LOCATIONS:
Locations (4):
- Medical Center Comac Medical EOOD, Sofia, Bulgaria
- Germany (3):
  - CRS Clinical-Research-Services Mannheim GmbH, Mannheim, Baden-Wurttemberg
  - Charité Research Organisation GmbH, Berlin
  - CTC North GmbH & Co. KG, Hamburg

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.